CLINICAL TRIAL: NCT02169102
Title: Effect of Low Power Laser in Pain Modulation During Irreversible Inflammation of Tooth Pulp
Brief Title: Effect of Low Power Laser in Tooth Pain Modulation Caused by Irreversible Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Karen Müller Ramalho, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 08509912.3.0000.0075
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Pulpitis; Acute Pain
Keywords: Low power laser; Pulpitis; Pain
MeSH Terms: conditions — Pulpitis; Acute Pain; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Other)
  Interventions: Other: No additional Intervention (control)
- Sham Laser (Sham Comparator)
  Interventions: Radiation: Sham Laser Irradiation
- Laser 1 (Experimental): Low Power Laser applied at 0.16 Joules/point. 2 points of laser irradiation
  Interventions: Radiation: Laser 1 (at 0,16 Joules/point of irradiation)
- Laser 2 (Experimental): Low Power Laser applied at 16 Joules/point. 2 points of laser irradiation
  Interventions: Radiation: Laser 2 (1,6 Joules/point of irradiation)

INTERVENTIONS:
Other: No additional Intervention (control) — No additional intervention previously to the urgency endodontic treatment (Control)
  Arms: Control
Radiation: Sham Laser Irradiation — Fifteen minutes previously the urgency endodontic treatment, sham laser irradiation was performed in the tooth with irreversible inflammation in pulp.
  Arms: Sham Laser
Radiation: Laser 1 (at 0,16 Joules/point of irradiation) — Fifteen minutes previously the urgency endodontic treatment, laser irradiation will be performed in the tooth with irreversible inflammation in pulp at 0,16 Joules/point at 2 points (perpendicularly to tooth crown and in periapex region)
  Arms: Laser 1
Radiation: Laser 2 (1,6 Joules/point of irradiation) — Fifteen minutes previously the urgency endodontic treatment, laser irradiation will be performed in the tooth with irreversible inflammation in pulp at 1,6 Joules/point at 2 points (perpendicularly to tooth crown and in periapex region)
  Arms: Laser 2

SUMMARY:
Anxiety, pain and discomfort are common stressful situations that occur during the dentistry practice, especially in the urgency endodontic practice. Studies have concluded that low intensity laser therapy is effective in treating pain. However, most studies have reported the low intensity laser therapy in chronic pain, few studies have shown its application on acute pain and none have evaluated the low intensity laser´s analgesic effect in acute pain of the pulp inflammation. Since the pulp tissue has the peculiar characteristic to be surrounded by dentin, in acute pulpits, the inflammatory reaction is more complicated than usual. Furthermore, during the inflammatory process, sometimes anesthesia is not always completely effective. Thus, this present study aims to evaluate whether previous therapy with low intensity laser could, by its analgesic effect, promote greater comfort especially to this type of patient. 60 patients with acute pulpits pain will be selected to this study (randomized and double-blinded) and they will be divided in 4 groups:

Group 1 ( n=15) - Control Group; Group 2 (n=15) - Laser 1: 780 nanometers (nm); 40 milliwatts (mW); 4 seconds per point; 0.16 Joules/point; total irradiated points: 02; Group 3 (n=15) - Laser 2: 780nm; 40 mW; 40 seconds per point; 1.6 Joules/point, total irradiated points: 02; Group 4 (n=15) - Placebo group - Sham Laser Irradiation.

The pain will be evaluated by a visual analogue scale (VAS) in 3 different times: initial pain, pain immediately after and 15 minutes after interventions (laser irradiation, or sham laser irradiation). After that, patients with acute pulp irreversible inflammation will be submitted to conventional endodontic urgency treatment. Data concerning the need of complimentary local anesthesia will be also taken into account. Data of different groups and times will be statistically compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute pain due to irreversible inflammation of the a vital pulp tooth

Exclusion Criteria:

* Non-Intact Pulp chamber
* Necrotic pulp

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2014-06 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Tooth pain modulation during irreversible pulp inflammation after low power laser irradiation | Immediately after low power laser irradiation and 15 minutes after low power laser irradiation
  Pain will be measured through VAS (Visual Analog Scale).

SECONDARY OUTCOMES:
Need of anesthetic supplementation during urgency endodontic treatment | 15 minutes
  15 minutes after low power laser irradiation, patients will be submitted to endodontic urgency treatment adopted in School of Dentistry of University of São Paulo. The need of local anesthetic supplementation will be observed between the patients

CONTACTS AND LOCATIONS:
Overall Officials: Larissa MP Souza, DDS, Study Chair — School of Dentistry - University of São Paulo; Carlos A Adde, PhD, Study Chair — School of Dentistry - University of São Paulo; Karen M Ramalho, PhD, Principal Investigator — School of Dentistry - University of São Paulo; Isabel P Tortamano, PhD, Principal Investigator — School of Dentistry - University of São Paulo; Carlos P Eduardo, PhD, Study Director — School of Dentistry - University of São Paulo; Rodney G Rocha, PhD, Study Director — School of Dentistry - University of São Paulo
Locations (1):
- School of Dentistry - University of São Paulo, São Paulo, São Paulo, Brazil